CLINICAL TRIAL: NCT03464058
Title: A Phase 1 Study to Determine the Single and Repeat Dose Pharmacokinetics, Food Effect, PPI Drug Interaction, Safety and Tolerability of Oral Prototype Formulations of BOS172767 in Healthy Subjects
Brief Title: Study to Determine the Single and Repeat Dose Pharmacokinetics, Food Effect, Proton Pump Inhibitor (PPI) Drug Interaction, Safety and Tolerability of Oral Prototype Formulations of BOS172767 in Healthy Subjects
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Boston Pharmaceuticals (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Triple | Purpose: Basic Science
Other Study IDs: BOS172767-01; 2017-004002-18 (EudraCT Number); QCL118174 (Other: Quotient Study Number)
Record Dates: First submitted 2018-03-07; First posted 2018-03-13 (Actual); Last update posted 2020-11-18 (Actual); Status verified 2020-11

CONDITIONS: Healthy Subjects
Keywords: Pharmacokinetics; Food Effect; Proton Pump Inhibitors; Drug Interaction; Oral Prototype Formulations
MeSH Terms: interventions — Rabeprazole

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Masking Description: Part 1 and 2 of the study are open-label and therefore blinding is not required. Part 3 of the study is double-blind.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (13):
- Part 1: Regimen A (Experimental): Participants will be treated with a BOS172767 200 milligram (mg) spray dried dispersion tablet (2 × 100 mg tablets) in the fasted state on Day 1.
  Interventions: Drug: BOS172767 tablets
- Part 1: Regimen B (Experimental): Participants will be treated with a BOS172767 200 mg lipid capsule (2 × 100 mg capsules) in the fasted state on Day 1.
  Interventions: Drug: BOS172767 liquid capsules
- Part 1: Regimen C (Experimental): Participants will be treated with a BOS172767 200 mg micronized capsule (2 × 100 mg capsules) in the fasted state on Day 1.
  Interventions: Drug: BOS172767 micronized capsules
- Part 1: Regimen D (Experimental): Participants will be treated with a BOS172767 200 mg immediate release reference capsule formulation (2 × 100 mg capsules) in the fasted state on Day 1.
  Interventions: Drug: BOS172767 immediate release capsules
- Part 1: Regimen E (Experimental): Participants will be treated with a selected dose of a prototype formulation of BOS172767 in the fasted state on Day 1.
  Interventions: Drug: BOS172767 tablets; Drug: BOS172767 liquid capsules; Drug: BOS172767 micronized capsules; Drug: BOS172767 immediate release capsules
- Part 1: Regimen F (Experimental): Participants will be treated with a selected dose of a prototype formulation of BOS172767 in the fed state on Day 1.
  Interventions: Drug: BOS172767 tablets; Drug: BOS172767 liquid capsules; Drug: BOS172767 micronized capsules; Drug: BOS172767 immediate release capsules
- Part 2: Regimen G (Experimental): Participants will be treated with 400 mg of the selected BOS172767 prototype in the fasted state on Day 1.
  Interventions: Drug: BOS172767 tablets; Drug: BOS172767 liquid capsules; Drug: BOS172767 micronized capsules; Drug: BOS172767 immediate release capsules
- Part 2: Regimen H (Experimental): Participants will be treated with 600 mg of the selected BOS172767 prototype in the fasted state on Day 1.
  Interventions: Drug: BOS172767 tablets; Drug: BOS172767 liquid capsules; Drug: BOS172767 micronized capsules; Drug: BOS172767 immediate release capsules
- Part 2: Regimen I (Experimental): Participants will be treated with 800 mg of the selected BOS172767 prototype in the fasted state on Day 1.
  Interventions: Drug: BOS172767 tablets; Drug: BOS172767 liquid capsules; Drug: BOS172767 micronized capsules; Drug: BOS172767 immediate release capsules
- Part 2: Regimen J (Experimental): Participants will be treated with rabeprazole on Days -3 to -1, and a selected dose of the BOS172767 prototype in the fasted state on Day 1.
  Interventions: Drug: BOS172767 tablets; Drug: BOS172767 liquid capsules; Drug: BOS172767 micronized capsules; Drug: BOS172767 immediate release capsules; Drug: Rabeprazole
- Part 3: Regimen K (Experimental): Participants will be treated with 400 mg of a BOS172767 prototype or matching placebo once daily (QD) or twice daily (BID) for 14 days (Days 1 to 14).
  Interventions: Drug: BOS172767 tablets; Drug: BOS172767 liquid capsules; Drug: BOS172767 micronized capsules; Drug: BOS172767 immediate release capsules; Drug: BOS172767 matching placebo capsules; Drug: BOS172767 matching placebo tablets
- Part 3: Regimen L (Experimental): Participants will be treated with 600 mg of a BOS172767 prototype or matching placebo QD or BID for 14 days (Days 1 to 14).
  Interventions: Drug: BOS172767 tablets; Drug: BOS172767 liquid capsules; Drug: BOS172767 micronized capsules; Drug: BOS172767 immediate release capsules; Drug: BOS172767 matching placebo capsules; Drug: BOS172767 matching placebo tablets
- Part 3: Regimen M (Experimental): Participants will be treated with 800 mg of a BOS172767 prototype or matching placebo QD or BID for 14 days (Days 1 to 14).
  Interventions: Drug: BOS172767 tablets; Drug: BOS172767 liquid capsules; Drug: BOS172767 micronized capsules; Drug: BOS172767 immediate release capsules; Drug: BOS172767 matching placebo capsules; Drug: BOS172767 matching placebo tablets

INTERVENTIONS:
Drug: BOS172767 tablets — Oral tablets
  Arms: Part 1: Regimen A; Part 1: Regimen E; Part 1: Regimen F; Part 2: Regimen G; Part 2: Regimen H; Part 2: Regimen I; Part 2: Regimen J; Part 3: Regimen K; Part 3: Regimen L; Part 3: Regimen M
Drug: BOS172767 liquid capsules — Oral capsules
  Arms: Part 1: Regimen B; Part 1: Regimen E; Part 1: Regimen F; Part 2: Regimen G; Part 2: Regimen H; Part 2: Regimen I; Part 2: Regimen J; Part 3: Regimen K; Part 3: Regimen L; Part 3: Regimen M
Drug: BOS172767 micronized capsules — Oral capsules
  Arms: Part 1: Regimen C; Part 1: Regimen E; Part 1: Regimen F; Part 2: Regimen G; Part 2: Regimen H; Part 2: Regimen I; Part 2: Regimen J; Part 3: Regimen K; Part 3: Regimen L; Part 3: Regimen M
Drug: BOS172767 immediate release capsules — Oral capsules
  Arms: Part 1: Regimen D; Part 1: Regimen E; Part 1: Regimen F; Part 2: Regimen G; Part 2: Regimen H; Part 2: Regimen I; Part 2: Regimen J; Part 3: Regimen K; Part 3: Regimen L; Part 3: Regimen M
Drug: BOS172767 matching placebo capsules — Oral capsules
  Arms: Part 3: Regimen K; Part 3: Regimen L; Part 3: Regimen M
Drug: BOS172767 matching placebo tablets — Oral tablets
  Arms: Part 3: Regimen K; Part 3: Regimen L; Part 3: Regimen M
Drug: Rabeprazole — Oral tablets
  Arms: Part 2: Regimen J

SUMMARY:
Part 1 of the study will be conducted to provide additional information on the safety and tolerability of single doses of BOS172767 in healthy participants, to evaluate the pharmacokinetic (PK) profiles (including relative bioavailability) of BOS172767 following oral administration of 3 prototype formulations in healthy participants compared to an immediate release capsule formulation (reference), and also to determine the relative bioavailability of a selected BOS172767 prototype formulation in the fed and fasted states.

Part 2 of the study will be conducted to provide additional information on the safety and tolerability of escalating single doses of the selected formulation of BOS172767 in healthy participants, to evaluate the PK profile following increased single doses of the selected formulation of BOS172767 following administration in healthy participants, and also to evaluate the dose linearity of the selected prototype.

Part 3 of the study will be conducted to provide additional information on the safety, tolerability, and PK of the selected formulation of BOS172767 following multiple ascending doses (MADs) over 14 days of dosing in healthy participants.

DETAILED DESCRIPTION:
Part 1 is comprised of a single-dose, part-randomized, open-label, 6-way crossover in 12 healthy participants. Participants will be dosed on 6 separate occasions (in 6 treatment periods), and will receive a single prototype of BOS172767 in each treatment period.

Part 2 is comprised of a single ascending dose, fixed-sequence, open-label, 3-way crossover with an optional fourth dosing period in 10 healthy participants. Participants will be dosed on 4 separate occasions (in 4 treatment periods), and will receive a single prototype of BOS172767 in each treatment period.

Part 3 is a double-blind (sponsor-open), placebo-controlled, randomized MAD part in 36 healthy participants (12 per study cohort). Participants will be dosed on 3 separate occasions (in 3 treatment periods), and will receive a single prototype of BOS172767 in each treatment period.

Parts 2 and 3 are contingent upon successful completion of Part 1.

ELIGIBILITY:
Inclusion Criteria:

* Healthy males or healthy females of non-child bearing potential
* Age 18 to 50 years of age at time of signing informed consent
* Body mass index of 18.0 to 32.0 kilograms per meters squared (kg/m^2) at Screening, or, if outside the range, considered not clinically significant by the investigator
* Must be willing and able to communicate and participate in the whole study
* Must have a negative Quantiferon tuberculosis test at Screening
* Must provide written informed consent
* Must agree to use an adequate method of contraception

Exclusion Criteria:

* Participants who have received any investigational medicinal product (IMP) in a clinical research study within the previous 3 months prior to dosing
* Participants who are study site employees, or immediate family members of a study site or sponsor employee
* Participants who have previously been enrolled (dosed) in this study
* History of any drug or alcohol abuse in the past 2 years prior to Screening
* Regular alcohol consumption in males >21 units per week and females >14 units per week (1 unit = ½ pint beer, 25 milliliters [mL] of 40% spirit or a 125 mL glass of wine)
* Current smokers and those who have smoked within the last 12 months prior to Screening. A breath carbon monoxide reading of greater than 20 parts per million at Screening or admission
* Current users of e-cigarettes and nicotine replacement products and those who have used these products within the last 12 months prior to Screening
* Females of childbearing potential
* Participants who do not have suitable veins for multiple venepunctures/cannulation as assessed by the investigator at Screening
* Clinically significant abnormal biochemistry, haematology or urinalysis as judged by the investigator
* Confirmed positive drugs of abuse test result
* Positive hepatitis B surface antigen, hepatitis C virus antibody or human immunodeficiency virus results
* Evidence of renal impairment at Screening, as indicated by an estimated creatinine clearance of <70 mL/minute using the Cockcroft-Gault equation
* History of clinically significant cardiovascular, renal, hepatic, chronic respiratory or gastrointestinal disease (including gall stones and/or cholecystectomy), neurological or psychiatric disorder, as judged by the investigator
* Serious adverse reaction or serious hypersensitivity to any drug or the IMP formulation excipients
* Adverse reaction to rabeprazole, its excipients or any proton pump inhibitors (Part 2 only)
* Presence or history of clinically significant allergy requiring treatment, as judged by the investigator. Hay fever is allowed unless it is active.
* Donation or loss of greater than 400 mL of blood within the previous 3 months
* Participants who are taking, or have taken, any prescribed or over-the-counter drug (other than 4 grams per day paracetamol or hormone replacement therapy) or herbal remedies in the 14 days before IMP administration. Exceptions may apply on a case by case basis, if considered not to interfere with the objectives of the study, as agreed by the Principal Investigator and sponsor's medical monitor.
* Participants who have any ongoing fungal infections (stable toe nail onychomycosis is allowed)
* Failure to satisfy the investigator of fitness to participate for any other reason

Ages: 18 Years to 50 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 28 (Actual)
Dates: Start 2018-03-21 (Actual); Primary Completion 2018-10-09 (Actual); Study Completion 2018-10-10 (Actual)

PRIMARY OUTCOMES:
Parts 1, 2, and 3: Number of participants with any treatment-emergent serious adverse event (TESAE) | up to 33 weeks
Parts 1, 2, and 3: Number of participants with any treatment-emergent non-serious adverse event (TEAE) | up to 33 weeks
Parts 1, 2, and 3: Number of participants with abnormal, clinically significant physical examination findings | up to 33 weeks
Parts 1, 2, and 3: Number of participants with abnormal, clinically significant safety laboratory test findings | up to 33 weeks
Parts 1, 2, and 3: Number of participants with abnormal, clinically significant vital sign values | up to 33 weeks
Parts 1, 2, and 3: Number of participants with abnormal, clinically significant electrocardiogram findings | up to 33 weeks
Parts 1 and 2: Plasma concentration of BOS172722 | predose; 0.5, 1, 2, 3, 4, 6, 8, 10, 12, 16 hours postdose (Day 1); 24 and 36 hours postdose (Day 2); 48 hours postdose (Day 3)
Part 2 (Regimen I): Plasma concentration of BOS172722 | admission to pre-dose (admission to dosing), 0 to 6 (Day 1), 6 to 12 (Day 1), 12 to 24 (Day 1), and 24 to 48 (Days 2 to 3) hours postdose
Part 3: Plasma concentration of BOS172722 | Days 1 and 7: pre-dose; 0.5, 1, 2, 3, 4, 6, 8, 10, 12, 16, and 24 hours postdose. Days 4, 6, 9, 11, and 12: pre-dose. Day 14: pre-dose; 0.5, 1, 2, 3, 4, 6, 8, 10, 12, 16, 24, 48, 72, 96, and 120 hours post-final dose
Part 3 (Regimen M): Plasma concentration of BOS172722 | admission to pre-dose on Day 1; 0 to 6, 6 to 12, and 12 to 24 hours postdose on Days 1, 7, and 14

CONTACTS AND LOCATIONS:
Locations (1):
- Quotient Sciences, Nottingham, United Kingdom